CLINICAL TRIAL: NCT02369458
Title: Phase II Trial of Mitomycin C in Patients With Incurable p16 Positive Oropharyngeal and p16 Negative Head and Neck Squamous Cell Carcinoma (HNSCC) Resistant to Standard Therapies
Brief Title: Mitomycin C in Patients With Incurable p16 Positive Oropharyngeal and p16 Negative Head and Neck Squamous Cell Carcinoma (HNSCC) Resistant to Standard Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201503060
Record Dates: First submitted 2015-02-16; First posted 2015-02-24 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma, Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Mitomycin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: p16+ OPSCC (Experimental): * Mitomycin C given on Day 1 every 5 weeks (each cycle is 5 weeks).
  * Pegfilgrastim will be given on Day 2 of each cycle (subcutaneous injection)
  Interventions: Drug: Mitomycin-C; Drug: Pegfilgrastim
- Cohort 2: p16- HNSCC (Experimental): * Mitomycin C given on Day 1 every 5 weeks (each cycle is 5 weeks).
  * Pegfilgrastim will be given on Day 2 of each cycle (subcutaneous injection)
  Interventions: Drug: Mitomycin-C; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Mitomycin-C
  Other Names: Mitosol; Mitomycin
Drug: Pegfilgrastim
  Other Names: •Neulasta®; GCSF

SUMMARY:
No agent is known to have efficacy in patients with incurable HNSCC that progressed with prior platin, 5-FU, cetuximab and taxane. Herein lies the unmet need to be addressed by this trial. Based on the preclinical and clinical data presented, the investigators propose that mitomycin C will have anti-tumor activity in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed incurable HNSCC of the oral cavity, oropharynx, larynx, hypopharynx, and/or Level 1-3 neck node with non-cutaneous SCC and unknown primary. "Incurable" is defined as metastatic disease or a local or regional recurrence in a previously irradiated site that is unresectable (or patient declines resection).
* Progression following platin and immunotherapy given for incurable disease.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam per RECIST 1.1.
* Tissue available (either initial diagnostic or recurrent tissue specimen) for p16 testing.
* At least 18 years of age.
* ECOG performance status ≤ 3
* Adequate hematologic, renal, and hepatic function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcl
  * Platelets ≥ 75,000/mcl
  * Total bilirubin ≤ 1.5 mg/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN, unless bone metastasis is present in the absence of liver metastasis
  * Creatinine below ULN (males 0.7-1.30 mg/dl; females 0.6-1.10 mg/dl) OR Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 1 month after completing treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Other active malignancy with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only, carcinoma in situ of the cervix, or synchronous H&N primaries.
* Currently receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 7 days of start of study treatment.
* Known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days prior to treatment.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to mitomycin C or other agents used in the study.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with the study drugs. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Oppelt, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort B: p16- HNSCC: * Mitomycin C given on Day 1 every 5 weeks (each cycle is 5 weeks).
  * Pegfilgrastim will be given on Day 2 of each cycle (subcutaneous injection)
Period: Overall Study
Arm/Group | Cohort A: p16+ OPSCC | Cohort B: p16- HNSCC
Started | 35 | 13
Completed | 34 | 13
Not Completed | 1 | 0
Not completed — Determined to be not eligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: p16+ OPSCC | Cohort B: p16- HNSCC | Total
Number analyzed (Participants) | 35 | 13 | 48
Age, Continuous [Median (Full Range); unit: years] | 61 [45 to 81] | 61 [54 to 68] | 61 [45 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 34 | 8 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 13 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 35 | 8 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 13 | 48

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (TRR)
Description: * TRR will be evaluated separately in p16- (HPV-unrelated) HNSCC patients and in p16+ (HPV positive) OPSCC patients using two optimal two-stage Simon designs. In both cases, the expected TRR is 10%. A TRR of 30% is considered a clinically significant increase.
  * RECIST 1.1 will be used for this outcome.
Time Frame: Approximately 6 months (median 5.6 months with full range of 0.1-33.7 months)
Population: One participant in each arm were not evaluable for tumor response rate.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: p16+ OPSCC | Cohort B: p16- HNSCC
Number analyzed (Participants) | 33 | 12
Participants | 3 | 0

2. Primary Outcome: Tumor Response Rate (TRR) for Participants Enrolled Post October 2020
Description: * TRR will be evaluated in p16+ (HPV positive) OPSCC HNSCC patients
  * RECIST 1.1 will be used for this outcome.
Time Frame: Approximately 6 months (median 4.0 months with full range of 0.5-12.0 months)
Population: Only participants enrolled post October 2020 are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: p16+ OPSCC | Cohort B: p16- HNSCC
Number analyzed (Participants) | 11 | 0
Participants | 0 |

3. Secondary Outcome: Progression-free Survival (PFS)
Description: * PFS is defined as the duration of time from start of treatment to time of first radiologic confirmation of progression or death, whichever occurs first.
  * Progressive disease per RECIST 1.1
    * Target lesions - At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
    * Non-target lesions - Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Approximately 6 months (median 5.6 months with full range of 0.1-33.7 months)
Population: One participant in each arm were not evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: p16+ OPSCC | Cohort B: p16- HNSCC
Number analyzed (Participants) | 33 | 12
months | 2.2 [1.6 to 3.4] | 2.1 [1.0 to 3.0]

4. Secondary Outcome: Number of Participants With Grade 3/4/5 Adverse Events
Description: -Using CTCAE Version 3.0
Time Frame: 28 days after completion of treatment (median length of follow-up was 96 days, full range of 3-463 days)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: p16+ OPSCC and Cohort B: p16- OPSCC: * Mitomycin C given on Day 1 every 5 weeks (each cycle is 5 weeks).
  * Pegfilgrastim will be given on Day 2 of each cycle (subcutaneous injection)
Arm/Group | Cohort A: p16+ OPSCC and Cohort B: p16- OPSCC
Number analyzed (Participants) | 47
Participants | 26

5. Secondary Outcome: Overall Survival (OS)
Description: -Defined as the date of first treatment to the date of death, last date alive, or date of patient withdrawal.
Time Frame: Through completion of follow-up (median length of follow-up Cohort A= 6.6 months IQR 2.7-12.0 months, median length of follow-up Cohort B=3.2 months IQR 1.5-9.4 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: p16+ OPSCC | Cohort B: p16- HNSCC
Number analyzed (Participants) | 34 | 13
months | 6.6 [3.5 to 9.9] | 3.2 [1.5 to 9.4]

6. Other Pre Specified Outcome: Quality of Life as Measured by the EORTC QLQ-C30
Description: -EORTC QLQ-C30: this has a total score, one general QOL, and one "within the last week" subscale, as well as a general health item and a single overall QOL item. This study does not use current empirical guidelines for the EORTC-QLQ-30 global score with the understanding that both the magnitude and variance of scores vary considerably from patient to patient, from one time point to another and by such factors as disease condition, age, and comorbidity. The participants can choose from 1-4 with 1 being Not At All and 4 being Very Much.
Time Frame: Baseline, every 5 weeks, and end of treatment (estimated at 6 months)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Quality of Life as Measured by the Cognitive Failures Questions (CFQ)
Description: -Cognitive Failures Questions (CFQ) - has 3 subscales describing perception, memory, and motor function. A change in 1 standard deviation will be considered a perceptible difference. The participants can choose a scale from 0-4 with 0 being Never and 4 being Very Often.
Time Frame: Baseline, every 5 weeks, and end of treatment (estimated at 6 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: -Adverse events were collected from start of treatment through 28 days following day of last treatment (median length of follow-up was 96 days, full range of 3-463 days). -Adverse events and all cause mortality were not collected separately by cohort.
Groups:
- Cohort A: p16+ OPSCC and Cohort B: p16- HNSCC: * Mitomycin C given on Day 1 every 5 weeks (each cycle is 5 weeks).
  * Pegfilgrastim will be given on Day 2 of each cycle (subcutaneous injection)
Arm/Group | Cohort A: p16+ OPSCC and Cohort B: p16- HNSCC
All-Cause Mortality (participants affected / at risk) | 47/47
Serious Adverse Events (participants affected / at risk) | 21/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: p16+ OPSCC and Cohort B: p16- HNSCC (N=47)
Injury to carotid artery (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Double vision (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Fever (General disorders) | 1
Pain (General disorders) | 1
Tumor fevers (General disorders) | 1
Device related infection (Infections and infestations) | 1
Infection with normal ANC - catheter related (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Midline shift (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: p16+ OPSCC and Cohort B: p16- HNSCC (N=47)
Anemia (Blood and lymphatic system disorders) | 45
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ear popping (Ear and labyrinth disorders) | 1
Hearing loss (no program) (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 3
Diabetes (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 16
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Salivary gland changes (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Xerostomia (Gastrointestinal disorders) | 9
Chills (General disorders) | 2
Edema: limb (General disorders) | 6
Edema: head and neck (General disorders) | 3
Fatigue (General disorders) | 29
Fever (General disorders) | 6
Hepatitis (drug induced suspected pembrolizumab) (Hepatobiliary disorders) | 1
Allergic reaction to CT dye (Immune system disorders) | 1
Allergic reaction to cetuximab (Immune system disorders) | 1
Allergic rhinitis (Immune system disorders) | 1
Infection with grade 3/4 neutrophils: upper airway (Infections and infestations) | 1
Infection with normal ANC: catheter (Infections and infestations) | 1
Infection with normal ANC: skin (Infections and infestations) | 1
Infection with normal ANC: tooth (Infections and infestations) | 1
Infection with normal ANC: upper airway NOS (Infections and infestations) | 6
Infection with normal ANC: chronic urinary tract infections (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 7
Creatinine increased (Investigations) | 8
INR increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 42
Neutrophil count decreased (Investigations) | 3
PTT increased (Investigations) | 2
Platelet count decreased (Investigations) | 19
Weight loss (Investigations) | 7
White blood cell count decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 1
High cholesterol (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 27
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 21
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Fracture - rib (Musculoskeletal and connective tissue disorders) | 1
Joint function (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Reflex sympathetic dystrophy (Musculoskeletal and connective tissue disorders) | 1
Rib pain (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 2
Hemorrhage, tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Accessory nerve disorder (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Sensory neuropathy (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 1
Benign prostatic hypertrophy (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal stones (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Acneiform rash (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Fingertip cracking (Skin and subcutaneous tissue disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Keratosis (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT02369458/Prot_SAP_001.pdf